CLINICAL TRIAL: NCT00939757
Title: A Phase 1, Open-Label, Randomized, Single Oral Dose, Three-Way Crossover Study to Assess the Effect of Food on the Pharmacokinetics of Mirabegron
Brief Title: Study of the Effect of Food on the Pharmacokinetics of Mirabegron
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 178-CL-041
Record Dates: First submitted 2009-07-13; First posted 2009-07-15 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-06

CONDITIONS: Healthy; Pharmacokinetics of Mirabegron
Keywords: Healthy volunteer subjects; pharmacokinetics; YM178; mirabegron; food
MeSH Terms: interventions — mirabegron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1. mirabegron, lower dose (Experimental)
  Interventions: Drug: mirabegron
- 2. mirabegron, higher dose (Experimental)
  Interventions: Drug: mirabegron

INTERVENTIONS:
Drug: mirabegron — oral tablet
  Other Names: YM178

SUMMARY:
The purpose of this study is to assess the effect of food on the pharmacokinetics of a single oral dose of mirabegron in healthy male and female subjects.

DETAILED DESCRIPTION:
Subjects will be assigned in a random order to receive 3 dosing regimens:

1. a single oral dose under a fasting condition;
2. a single oral dose with food (low fat breakfast);
3. a single oral dose with food (high fat breakfast).

ELIGIBILITY:
Inclusion Criteria:

* The subject must weigh at least 45 kg and have a body mass index (BMI) between 20.0 and 32.0 kg/m2 , inclusive
* The subject must have a normal or clinically non-significant 12 lead ECG as well as normal or clinically non-significant laboratory test results
* Female subjects must be post-menopausal (defined as at least 2 years without menses), surgically sterile, or practicing effective contraception, and will continue to use effective contraception during the study period. All females must be non-lactating, and must have a negative pregnancy test result
* The subject must have negative test results for drugs of abuse and alcohol screens
* The subject must have good venous access in both arms

Exclusion Criteria:

* The subject has evidence of QTc interval >430 msec for male, >450 msec for female
* The subject has liver function test values (ALT, AST, or bilirubin) above the upper limit of normal
* The subject has a history or presence of psychiatric illness, serious active or recurrent infection, or any medical condition or disorder that precludes the subject from participating in the study
* The subject has a previous history of cancer other than basal cell carcinoma or Stage 1 squamous cell carcinoma that has not been in remission for at least 5 years
* The subject has donated or lost ≥ 450 mL blood within 56 days prior to study drug administration or has donated plasma within 7 days prior to study drug administration
* The subject has received or is anticipated to receive a prescription drug within 14 days prior to Day -1 of Period 1 (within 30 days 1 for any long acting treatments such as depot formulations). Subject has taken any over-the-counter (OTC) medications, including complementary and alternative medicines (except for oral contraceptives and occasional use of acetaminophen of up to 2000 mg/day but not more than 4 days per week) within 14 days
* The subject has consumed alcohol, xanthine derivative-containing food/beverages (tea, chocolate), grapefruit juice, grapefruit-containing products or Seville oranges (e.g., bitter marmalade) within 48 hours before admission into the unit
* The subject has used tobacco-containing products and nicotine-containing products within 6 months
* The subject consumes more than 5 units of alcoholic beverages (one unit is 12 ounces of beer, 4 ounces of wine or 1 ounce of spirits) per week, or has a history of substance abuse, drug addiction, or alcoholism within past 2 years
* The subject is known to have hepatitis or HIV-1 and/or HIV-2, or is positive for hepatitis A antibody IgM, hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2009-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Assess the effects of food on the pharmacokinetics of a single oral dose of mirabegron | 4-5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Global Development
Locations (1):
- Tacoma, Washington, United States

REFERENCES:
- [Background] Lee J, Zhang W, Moy S, Kowalski D, Kerbusch V, van Gelderen M, Sawamoto T, Grunenberg N, Keirns J. Effects of food intake on the pharmacokinetic properties of mirabegron oral controlled-absorption system: a single-dose, randomized, crossover study in healthy adults. Clin Ther. 2013 Mar;35(3):333-41. doi: 10.1016/j.clinthera.2013.02.014. PMID 23497763